CLINICAL TRIAL: NCT00811681
Title: Effect of Pioglitazone Administered to Patients With Friedreich's ATAXIA:Proof of Concept
Brief Title: Effect of Pioglitazone Administered to Patients With Friedreich's Ataxia: Proof of Concept
Acronym: ACTFRIE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P070123
Record Dates: First submitted 2008-12-18; First posted 2008-12-19 (Estimated); Last update posted 2013-09-04 (Estimated); Status verified 2013-08

CONDITIONS: Friedreich's Ataxia
Keywords: Friedreich's ataxia; Pioglitazone
MeSH Terms: conditions — Friedreich Ataxia | interventions — Pioglitazone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pioglitazone (Experimental): pioglitazone
  Interventions: Drug: pioglitazone
- Control (Placebo Comparator): placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: pioglitazone — administered orally once a day after the first visit and for a total of 2 years. Initially, Pioglitazone will be started at 15mg /day. Dosage will then increase by 15mg /d/ week up to the maximal dose of 45mg /day
  Arms: Pioglitazone
Drug: Placebo — a placebo administered orally once a day after the first visit and for a total of 2 years.
  Other Names: Control
  Arms: Control

SUMMARY:
Friedreich's ataxia (FA) is a rare progressive neurological disorder affecting approximately 1/30, 000 individuals. No treatment is presently available to counteract the neurodegeneration of this extremely severe disease.

Pioglitazone, a well known PPAR gamma (peroxysome proliferators-activated receptor gamma) ligand induces the expression of many enzymes involved in the mitochondrial metabolism, including the superoxide dismutases. This agent may be therapeutic by counteracting the disabled recruitment of antioxidant enzymes in FA patients. This potential neuroprotective agent crosses the brain blood barrier in human.

Primary objective: To explore the effects of Pioglitazone on neurological function in FA patients. We expect neurological benefits taking into account the natural course of the disease.

Population: Subjects for this study will be limited to patients not older than 25 years Methodology: Prospective, randomized double-blind trial of Pioglitazone versus placebo in FA patients. Patients will be treated two years and will undergo clinical exams and testing during three days each six months at the clinical investigation centre.

DETAILED DESCRIPTION:
State of the art Friedreich's ataxia (FA) is a rare progressive neurological disorder affecting approximately 1/30, 000 individuals. No treatment is presently available to counteract the neurodegeneration of this extremely severe disease. The cardinal feature is a progressive gait and limb ataxia. Other commonly associated clinical signs include: dysarthria, sensory loss, distal weakness, pyramidal signs, absent reflexes, nystagmus and cardiomyopathy. Pes caves, scoliosis, diabetes and decline of vision or audition are also found in many patients. The disease often reveals before adulthood and leads to a progressive loss of autonomy about ten years after disease onset. FA is recessively inherited with a GAA trinucleotide repeat expansion in the first intron of a gene encoding frataxin a mitochondrial protein. Decreased frataxin leads to a mitochondrial iron-sulfur protein deficiency and hampered signalling pathways for superoxide dismutases, key enzymes of early antioxidant defences of the cells. As a result, cultured patient cells are particularly sensitive to oxidative insult. One aspect of the pathogenesis in vivo might be explained by this phenomenon.

Pioglitazone, a well known PPAR gamma (peroxysome proliferators-activated receptor gamma) ligand induces the expression of many enzymes involved in the mitochondrial metabolism, including the superoxide dismutases. This agent may be therapeutic by counteracting the disabled recruitment of antioxidant enzymes in FA patients. This potential neuroprotective agent crosses the brain blood barrier in human. A clinical study has shown that a daily treatment with Pioglitazone during three years induced apparent clinical improvement without adverse events in multiple sclerosis patients. Pioglitazone has been shown to possibly act on neurodegeneration in humans and animals models thus it appears a promising agent to be tested in Friedreich ataxia. This agent also didn't show any peculiar toxicity in cultured human cells with low frataxin compared with control. All these facts lead us to propose a clinical trial with Pioglitazone in patients with FA. .

Primary objective: To explore the effects of Pioglitazone on neurological function in FA patients. We expect neurological benefits taking into account the natural course of the disease.

Population: Subjects for this study will be limited to patients not older than 25 years Methodology: Prospective, randomized double-blind trial of Pioglitazone versus placebo in FA patients. Patients will be treated two years and will undergo clinical exams and testing during three days each six months at the clinical investigation centre.

Patients number justification: 20 patients in each group will be enrolled in the study with considerations to inclusion possibilities and the Bayes statistical analysis methodology. Evaluation of prior distribution of success probability per arm will be based on previous literature data and experts consensus.

Primary endpoint : change in neurological testing as performed using the International Cooperative Ataxia Rating Scale (ICARS) settled down by the World Federation of Neurology. Success will be defined as a stabilisation or improvement on ICARS designed as no more than 2 points maximum increment on this scale in two years.

Secondary endpoints include measurements of the following: Neurological score by the Friedreich's Ataxia Rating Scale (FARS), gait record and analysis of its components, posture study, kinetic study of the upper limbs, speech, oculomotor and auditory disorders, functional handicap using the Disability Status Scale (DSS), quality of life by SF-36 score; Cardiac involvement (electrocardiography, 24 hours holter, echocardiography with tissue doppler) and drug tolerance.

Benefits expected with this clinical trial: Expected results will be reduced symptoms or stabilization of the natural evolution of this threat full progressive disease with bad prognosis in patients treated with Pioglitazone. Furthermore, study results will possibly contribute in the validation and standardization of new clinical evaluation tools used in the follow-up of Friedreich ataxia patients.

Specific monitoring was initiated in all patients included in the study taking into account a potential risk of bladder cancer.

All patients included in the protocol ACTFRIE, will be asked to participate in the study of tolerance. They will receive pioglitazone at a dose of 45 mg per day, until the data on the effectiveness or otherwise of this treatment, its side effects in patients with Friedreich's ataxia are known by the results of ACTFRIE testing (approximately April 2014).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of FA with confirmed FRDA mutations
* GAA repeat length of the shorter allele of frataxin gene > 300
* Age ≤ 24 years
* Ambulatory (assistance devices permitted) or able to stand up without support
* Neurologically symptomatic
* All subjects agree and commit to the use of 2 reliable methods of birth control for the duration of the study if sexually active
* Willing (and parents if minor) to participate in all aspects of trial design and follow-up
* No modification of the usual treatment 6 months before inclusion and agree to stay with the same treatment during the trial (idebenone with a stable dosage, cardiologic therapeutic)

Exclusion Criteria:

* Composite heterozygote
* Patients unable to stand up even with support
* Pregnant women
* Cardiac insufficiency NYHA III to IV and heart ejection fraction> 50%
* Alkaline phosphatase, SGOT or SGPT greater than 1.5 X the upper limit of normal
* Patients with diabetes
* Modification of the concomitant medications taken by the patient within the 6 months before inclusion or during the trial
* Clinically significant medical disease that, in the judgment of the investigators, would expose the patient to undue risk of harm or prevent the patient from completing the study.

Ages: 7 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2008-12; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
evaluate the efficacy of Pioglitazone on the neurological function of FA patients. Success will be defined as a stabilisation or improvement on ICARS designed as no more than 2 points maximum increment on this scale in two year. | 2 years

SECONDARY OUTCOMES:
tolerance of Pioglitazone | 2 years
efficacy of Pioglitazone on neurological function | 2 years
efficacy of Pioglitazone on functional handicap and quality of life | 2 years
effect of Pioglitazone on cardiac parameters | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Husson, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Robert Debré, Paris, France

REFERENCES:
- [Derived] Simon AL, Meyblum J, Roche B, Vidal C, Mazda K, Husson I, Ilharreborde B. Scoliosis in Patients With Friedreich Ataxia: Results of a Consecutive Prospective Series. Spine Deform. 2019 Sep;7(5):812-821. doi: 10.1016/j.jspd.2019.02.005. PMID 31495483